CLINICAL TRIAL: NCT06712420
Title: Neoadjuvant Chemotherapy Versus Upfront Surgery for Locally Advanced Resectable Gall Bladder Cancer : A Randomized Trial
Brief Title: Neoadjuvant Chemotherapy for Locally Advanced Gall Bladder Cancer : a Randomized Control Trial (NEOGB)
Acronym: NEOGB
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Rajiv Gandhi Cancer Institute & Research Center, India (Other)
Responsible Party: Principal Investigator, Shaifali Goel, DOCTOR, Rajiv Gandhi Cancer Institute & Research Center, India
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RGCIRC/IRB-BHR/26/2024; RES/SCM/61/2023/89 (Other: RAJIV GANDHI CANCER INSTITUTE AND REASEARCH CENTRE,INDIA)
Record Dates: First submitted 2024-10-22; First posted 2024-12-02 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Gall Bladder Carcinoma
Keywords: gallbladder, locally advanced, neoadjuvant
MeSH Terms: conditions — Gallbladder Neoplasms | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- upfront surgery (Experimental): after staging workup and biopsy, patient being taken up for upfront surgical exploration will undergo staging laparoscopy followed by exploration and interaortocaval lymphnode sampling. After ruling out distant metastasis, local resectability will be reassessed and curative surgery will be performed. . Post-operative complications were recorded and graded according Clavien Dindo classification
  Interventions: Procedure: curative surgery
- Neoadjuvant chemotherapy followed by surgery (Experimental): NACT group will receive gemcitabine and platinum combination. Most common regimen comprised of gemcitabine (1000 mg/ m2 intravenously over 30-60 min) on days 1 and 8, and cisplatin (75 mg/ m2 intravenously over 2 h) on day 1, every 21 days. In case of renal compromise, carboplatin was used. Response was assessed using CECT abdomen and PET scan. Chemotherapy related toxicity will be graded according to Common Terminology Criteria for Adverse Events (CTCAE) v 5 .0.
  Interventions: Drug: neoadjuvant chemotherapy; Procedure: curative surgery

INTERVENTIONS:
Drug: neoadjuvant chemotherapy — NACT group will receive gemcitabine and platinum combination. Most common regimen comprised of gemcitabine (1000 mg/ m2 intravenously over 30-60 min) on days 1 and 8, and cisplatin (75 mg/ m2 intravenously over 2 h) on day 1, every 21 days. In case of renal compromise, carboplatin was used. Response was assessed using CECT abdomen and PET scan. Chemotherapy related toxicity will be graded according to Common Terminology Criteria for Adverse Events (CTCAE) v 5 .0. PAtients will undergo curative surgery after neoadjuvant chemotherapy
  Other Names: NACT
  Arms: Neoadjuvant chemotherapy followed by surgery
Procedure: curative surgery — Patient being taken up for surgical exploration will undergo staging laparoscopy followed by exploration and interaortocaval lymphnode sampling. After ruling out distant metastasis, local resectability will be reassessed and curative surgery will be performed. . Post-operative complications were recorded and graded according Clavien Dindo classification

SUMMARY:
to study role of chemotherapy treatment for gall bladder cancer before surgery as compared to surgery directly

DETAILED DESCRIPTION:
Gallbladder cancer is a highly aggressive disease with a late presentation and poor prognosis. Complete surgical excision remains the only potentially curative treatment for early-stage gallbladder cancer.

The use and benefit of chemotherapy in gallbladder cancer before surgery , that is , in the neoadjuvant setting, is not well studied and, to our knowledge, neoadjuvant chemotherapy has not been evaluated in any randomized clinical trial.

Neoadjuvant chemotherapy aims to achieve tumor downstaging, increase the radical surgical resection rate, reduce metastases. This study will compare the effectiveness of chemotherapy before surgery in locally advanced gall bladder cancer versus upfront surgery with respect to survival and completeness of resection of disease.

ELIGIBILITY:
Inclusion Criteria:

* ECOG 0-2
* Locally advanced resectable GBC defined as Clinical T3/4 disease or Regional LN involvement on imaging studies.
* Post cholecystectomy GBC with residual disease on imaging, History of bile spillage during primary surgery , history of piece-meal removal of gall bladder during simple cholecystectomy, Regional LN involvement on imaging studies.

Exclusion Criteria:

1. Early GBC ( cT1/T2) without significant lymphadenopathy or liver infiltration on radiological imaging .
2. Locally advanced disease requiring major hepatectomy or whipple's pancreatoduodenectomy.
3. Post cholecystectomy GBC without any evidence of spillage of residual disease on radiological imaging.
4. Obstructive jaundice due to involvement of biliary tree by tumour.
5. Vascular involvement such as common hepatic artery, MPV right hepatic artery or right portal vein.
6. Any distant metastasis or isolated port site metastasis
7. Involvement of non-regional LN (e.g . Celiac LN, SMA lymph node, inter-aortocaval or left para-ortic LN).
8. Poor performance status ECOG 3 or more.
9. Pregnancy.
10. Inability or unwillingness to follow study protocol

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
improvement in 3 year overall survival | 3 year
  To compare the 3 year overall survival with Neoadjuvant chemotherapy and surgery versus upfront surgery in locally advanced resectable gall bladder cancer

SECONDARY OUTCOMES:
post operative outcomes | 90 days
  To compare mortality and morbidity rate in two groups

CONTACTS AND LOCATIONS:
Overall Officials: Shivendra Singh, Mch Surgical gastroenterology, Study Director — Rajiv Gandhi Cancer Institute and Research Centre
Locations (1):
- Rajiv Gandhi Cancer Institute and Research Centre, Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No
Institutional Policy